CLINICAL TRIAL: NCT01991951
Title: Prospective Randomized Study of Incidence of Thromboembolic and Bleeding Events According to the Period of Warfarin Use Before and After Catheter Ablation of Paroxysmal Atrial Fibrillation in Low Risk Patients
Brief Title: Short Term Warfarin Therapy for Radiofrequency Catheter Ablation of Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Young-Hoon Kim, Professor of medicine, Korea University Anam Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUMCEP01
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin

ARMS (2):
- Short term warfarin group (Experimental): taking warfarin for only 2 weeks after catheter ablation of atrial fibrillation
  Interventions: Drug: warfarin
- Conventional therapy arm (Active Comparator): conventional warfarin therapy of 3 weeks before and 8 weeks after catheter ablation of AF
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: warfarin

SUMMARY:
We hypothesized that in patients with low CHADS-VASc score (2 or < 2), there is no difference in thromboembolic or bleeding events between patients with short term warfarin therapy (2 weeks after catheter ablation) and conventional therapy (3 weeks before and 8 weeks after procedure).

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal atrial fibrillation who underwent radiofrequency catheter ablation
* Patients with CHADS-VASc score 2 or less than 2

Exclusion Criteria:

* Patients who do not consent to the study
* Permanent or persistent atrial fibrillation
* Patients who have underwent prior catheter ablation for atrial fibrillation
* CHADS-VASc score more than 2
* History of stroke
* LVEF <40%
* Significant liver or kidney dysfunction
* History of major bleeding during warfarin therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of thromboembolic and bleeding events during 2 months | 2 months after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea